CLINICAL TRIAL: NCT02609347
Title: Immediate Effects of Manual Therapy for Patients After Ankle/Hindfoot Fractures
Brief Title: Manual Therapy After Ankle/Hindfoot Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Stephanie Albin, DPT, OCS, FAAOMPT, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1050061
Record Dates: First submitted 2015-10-29; First posted 2015-11-20 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Ankle Fracture; Calcaneus Fracture; Talus Fracture; Pilon Fracture
Keywords: Manual Therapy; Ankle Fracture; Hindfoot Fracture
MeSH Terms: conditions — Ankle Fractures | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy Group (Experimental): Participants in the manual therapy group will receive 3 treatment sessions of joint mobilization based on the physical therapist's clinical decision making.
  Interventions: Other: Manual Therapy Group
- Control Group (Sham Comparator): Participants in the control group will receive a sham manual therapy treatment consisting of soft tissue mobilization and Grade I mobilizations at the proximal tib/fib joint.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Manual Therapy Group — The manual therapy intervention will be based on the typed of fracture the patient sustained, and their limitations in joint mobility.
  Arms: Manual Therapy Group
Other: Control Group — The sham intervention will consist of soft tissue mobilization and Grade I mobilization at the proximal tib/fib joint.
  Arms: Control Group

SUMMARY:
The aim of this randomized controlled trial is to assess if manual therapy improves mobility, gait, and balance more than a control group for patients who have undergone open reduction internal fixation (ORIF) after an ankle/hindfoot fracture.

DETAILED DESCRIPTION:
This study will enroll 76 subjects with stiffness after ankle and/or hindfoot fractures. Stiffness will be defined in this study with the ankle lunge test. This test measures dorsiflexion (DF) in a weight bearing position, and a side-to-side difference of > 5.0 centimeters (cm) will be used for the criteria to determine ankle stiffness as this is greater than three times the smallest real difference of 1.38 cm. Potential subjects will be recruited by either their orthopedic surgeon or the PI and must satisfy all inclusion/exclusion criteria. Those individuals meeting the eligibility criteria who agree to participate and sign an informed consent from the appropriate Internal Review Board (IRB) will undergo a baseline assessment. The baseline assessment will be performed by a clinician blinded to the subject's treatment group assignment. Participants will be randomized to receive manual therapy (MT) or to the control group (CONTROL) based on a list generated by a computer program and sequentially numbered and placed in a sealed envelope after baseline measures are completed. Participants will then be given a chance to practice the functional tests prior to the baseline assessment, and will have a chance to rest if needed. The order in which tests are administered will be randomized by a computer generated process. Participants will be asked to perform the following tests: single limb stance (average of 3 trials), the Star excursion balance test (anterior, posteromedial, and posterolateral directions only) (average of 3 trials), the ankle lunge test (ALT), the foot assessment platform, the MyotonPRO and walk across the GAITRite mat. Patients will perform all tests without shoes in order to standardize footwear between subjects, and all tests will be performed on both the affected and unaffected sides.

After all baseline measures have been taken, participants will be randomized to either the MT or the Control Group. Participants in the manual therapy group will receive joint mobilization and participants in the control group will receive a sham manual therapy treatment consisting of soft tissue mobilization and Grade I mobilizations at the proximal tib/fib joint. Treatment for the manual therapy group will be based on the physical therapist's clinical decision making that is fellowship trained in manual therapy. For instance, if a patient has a talar neck fracture and is lacking dorsiflexion, the therapist may choose to avoid an anterior-posterior talocrural joint mobilization which may place increased stress through the talar neck and mobilize instead the talonavicular joint and/or the subtalar joint based on stiffness.

After receiving treatment, participants will again perform the tests and measures in a random order, and will be allowed to rest as much as needed. The amount of time needed to rest between tests will be documented. Participants will return for 2 additional follow up visits between 7 to 10 days after the initial examination and measurements; however, they will only be asked to fill out the self-reported questionnaires and perform the tests and measures after the second treatment. Participants will then follow up between 7-10 days after their last manual therapy treatment for a final measurement of all tests and measures. Participants in the control group will be asked to follow-up at the same time points as the manual therapy group after their initial baseline measures and asked to complete all questionnaires and tests at the same time points as the manual therapy group. Subjects will be asked to avoid practicing balance and beginning exercises other than normal activities of daily living during this time.

Specific Aim 1: To evaluate if manual therapy improves range of motion, muscle stiffness, and in patients with ankle stiffness after ankle/hindfoot fractures more than a control group.

The dependent variables for Aim1 are weight bearing dorsiflexion range of motion (ROM), foot mobility, and muscle stiffness. The independent variables for Aim1 are treatment group (MT vs CONTROL) and time. The primary aim will be examined using a linear mixed model with repeated measures to account for the correlation among repeated observations from the same patient. Time (baseline, assessment 1 and assessment 2) and treatment group (MT and CONTROL) will be modeled as fixed effects, with the ALT as the primary dependent variable (DV). Separate models will be constructed in a similar fashion with foot mobility magnitude (FMM) and muscle stiffness as the DV. The hypothesis of interest will be the group-by-time interaction. Treatment effects will be calculated from the between-group differences in change score from baseline to assessment 1 and assessment 2.

Specific Aim 2: To evaluate if patients receiving three manual therapy treatments will have greater improvements in spatial and temporal gait parameters than a control group.

The dependent variables for Aim 2 are gait velocity and stance times. The independent variables for Aim 2 are treatment group (MT vs CONTROL) and time. The primary aim will be examined using a linear mixed model with repeated measures to account for the correlation among repeated observations from the same patient. Time (baseline, assessment 1 and assessment 2) and treatment group (MT and CONTROL) will be modeled as fixed effects, with gait velocity as the primary dependent variable (DV). A separate model will be constructed in a similar fashion with stance time as the DV. The hypothesis of interest will be the group-by-time interaction. Treatment effects will be calculated from the between-group differences in change score from baseline to assessment 1 and assessment 2.

Specific Aim 3: To evaluate if patients receiving three manual therapy treatments will have greater improvement in balance than a control group.

The dependent variables for Aim3 are distances reached on the star excursion balance test and single limb stance times. The independent variables for Aim3 are treatment group (MT vs CONTROL) and time. The primary aim will be examined using a linear mixed model with repeated measures to account for the correlation among repeated observations from the same patient. Time (baseline, assessment 1 and assessment 2) and treatment group (MT and Control) will be modeled as fixed effects, with distance reached for the star excursion balance test (SEBT) as the primary dependent variable (DV). A separate model will be constructed in a similar fashion with single limb stance time as the DV. The hypothesis of interest will be the group-by-time interaction. Treatment effects will be calculated from the between-group differences in change score from baseline to assessment 1 and assessment 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Stiffness > 5.0 cm side to side difference as measured by the ankle lunge test
3. Surgical management of ankle or hindfoot fracture
4. Full weight-bearing (WB)
5. Able to read and speak sufficient English to complete outcome tools

Exclusion Criteria:

1. Any prior foot/ankle surgery, deformity, or injury on the unaffected side which would affect gait, WB dorsiflexion or balance
2. Unable to attend follow-up visits
3. Any cognitive impairments which would prevents patients from being able to complete or understand questionnaires
4. Have received any previous manual therapy for their current ankle and/or hindfoot fracture
5. Have a known non/malunion
6. Have additional fractures of the spine, hip, or knee that would likely affect their weight bearing or gait
7. Have avascular necrosis as demonstrated on radiographs
8. Syndesmotic screw intact
9. Open reduction internal fixation >12 months previously

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Range of motion (ROM) | 2 weeks
  The dependent variable for Aim1 is weight bearing dorsiflexion ROM. The independent variables for Aim1 are treatment group (Manual therapy group versus Control group) and time
Spatial and temporal gait parameters - gait velocity | 2 weeks
  The dependent variable for Aim 2 is gait velocity. The independent variables for Aim 2 are treatment group (Manual therapy group versus Control group) and time.
Balance | 2 weeks
  The dependent variables for Aim3 is distances reached on the star excursion balance test. The independent variables for Aim3 are treatment group (Manual therapy group versus Control group) and time.

SECONDARY OUTCOMES:
Characteristics that predict outcomes | 2 weeks
  Multiple linear regression analysis will be performed to determine if baseline characteristics such as fracture type, age, etc can predict changes in biomechanical outcomes
Foot Mobility - Foot Assessment Platform (FAP) | 2 weeks
  The dependent variable is foot mobility. The independent variables are treatment group (Manual therapy group versus Control group) and time. Foot mobility will be assessed using the FAP.
Muscle Stiffness - MyotonPRO Device | 2 weeks
  The dependent variable is muscle stiffness. The independent variables are group and time. Muscles stiffness will be assessed using the MyotonPRO device.
Stance Time | 2 weeks
  The dependent variable is stance time. The independent variables are group and time.
Single Limb Stance Time | 2 weeks
  The dependent variable is single limb stance time. The independent variables are treatment group (Manual therapy group versus Control group) and time.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie R Albin, DPT, FAAOMPT, Principal Investigator — Intermountain Health Care
Locations (1):
- Intermountain Healthcare, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Not planning on sharing data

REFERENCES:
- [Result] van Tetering EA, Buckley RE. Functional outcome (SF-36) of patients with displaced calcaneal fractures compared to SF-36 normative data. Foot Ankle Int. 2004 Oct;25(10):733-8. doi: 10.1177/107110070402501007. PMID 15566705
- [Result] Griffin D, Parsons N, Shaw E, Kulikov Y, Hutchinson C, Thorogood M, Lamb SE; UK Heel Fracture Trial Investigators. Operative versus non-operative treatment for closed, displaced, intra-articular fractures of the calcaneus: randomised controlled trial. BMJ. 2014 Jul 24;349:g4483. doi: 10.1136/bmj.g4483. PMID 25059747
- [Result] Balazs GC, Polfer EM, Brelin AM, Gordon WT. High seas to high explosives: the evolution of calcaneus fracture management in the military. Mil Med. 2014 Nov;179(11):1228-35. doi: 10.7205/MILMED-D-14-00156. PMID 25373046
- [Result] Schulze W, Richter J, Russe O, Ingelfinger P, Muhr G. Surgical treatment of talus fractures: a retrospective study of 80 cases followed for 1-15 years. Acta Orthop Scand. 2002 Jun;73(3):344-51. doi: 10.1080/000164702320155374. PMID 12143985
- [Result] Hirschmuller A, Konstantinidis L, Baur H, Muller S, Mehlhorn A, Kontermann J, Grosse U, Sudkamp NP, Helwig P. Do changes in dynamic plantar pressure distribution, strength capacity and postural control after intra-articular calcaneal fracture correlate with clinical and radiological outcome? Injury. 2011 Oct;42(10):1135-43. doi: 10.1016/j.injury.2010.09.040. Epub 2010 Nov 13. PMID 21075372
- [Result] O'Brien J, Buckley R, McCormack R, Pate G, Leighton R, Petrie D, Galpin R. Personal gait satisfaction after displaced intraarticular calcaneal fractures: a 2-8 year followup. Foot Ankle Int. 2004 Sep;25(9):657-65. doi: 10.1177/107110070402500911. PMID 15563389
- [Result] Simondson D, Brock K, Cotton S. Reliability and smallest real difference of the ankle lunge test post ankle fracture. Man Ther. 2012 Feb;17(1):34-8. doi: 10.1016/j.math.2011.08.004. Epub 2011 Sep 29. PMID 21959254
- [Result] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143
- [Result] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Result] McPoil TG, Vicenzino B, Cornwall MW, Collins N, Warren M. Reliability and normative values for the foot mobility magnitude: a composite measure of vertical and medial-lateral mobility of the midfoot. J Foot Ankle Res. 2009 Mar 6;2:6. doi: 10.1186/1757-1146-2-6. PMID 19267907